CLINICAL TRIAL: NCT01574352
Title: The Odense Overweight Intervention Study (OOIS): A Randomized Controlled Trial on Overweight Prevention in Children.
Brief Title: The Odense Overweight Intervention Study
Acronym: OOIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Southern Denmark (Other)
Collaborators: TrygFonden, Denmark (Industry)
Responsible Party: Principal Investigator, Lars Bo Andersen, Professor, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: S20120015
Record Dates: First submitted 2012-03-26; First posted 2012-04-10 (Estimated); Results first posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Children; Overweight; Obesity; Metabolic Syndrome
Keywords: Children; Overweight; Obesity; BMI; Physical activity; Cognitive function; Intervention study; Randomized controlled trial; Day camp; Risk factors
MeSH Terms: conditions — Overweight; Obesity; Metabolic Syndrome; Motor Activity | interventions — Control Groups; Behavior Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention camp (Experimental): Children's behavior are controlled each week day for six weeks, and children participate in three hours of physical activity every day
  Interventions: Behavioral: Intervention camp
- Small intervention (Experimental): Children are only informed of healthy behavior
  Interventions: Behavioral: Small intervention

INTERVENTIONS:
Behavioral: Small intervention — The control group are offered a weekly 1 hour training or activity session during six weeks. Furthermore two sessions where the parents are invited to participate in information about diet and exercise.
  Other Names: control group
  Arms: Small intervention
Behavioral: Intervention camp — The children are participating in a 6 week day camp. The camp contains social activities, physical activity training, usual school classes and health education. All meals (healthy food) are consumed during the camp day.
  Other Names: Behavioral intervention; Camp intervention; Physical activity intervention
  Arms: Intervention camp

SUMMARY:
Strong and consistent evidence have shown that overweight, including obesity, is an important risk factor for the development of cardiovascular disease (CVD) in adults. Several studies have found an association between overweight in childhood and increased risk of morbidity and mortality later in life. The prevalence of overweight in children and adolescents has increased in recent years, and consequently it is important to identify effective approaches in the prevention and treatment of overweight in young individuals.

Approaches such as resident weight loss camps have shown promising results. A residential camp setting provides an opportunity to increase and control exposure to, for instance, particular foodstuffs, beverages and physical activity opportunities. However, well-designed studies with sufficient participants are still needed on the reversal of overweight in childhood with increased focus on documenting predictors of behavior changes associated with decreases in overweight.

This study is carried through as a randomized controlled trial which investigates the effect of participating in a 6 week health promoting resident for overweight fifth grade children camp followed by 46 weeks of family support.

The study hypothesis is that participating in a 6 week resident camp and a following period of 46 weeks of child and family support will induce a reduction in body mass index (BMI). In addition it is expected that the intensity and duration intervention program is sufficient to cause changes in physiological parameters related to a reduced risk of lifestyle diseases.

DETAILED DESCRIPTION:
Intervention type 1: Day camp and resident camp:

The intervention is divided into two parts - an intensive six week day or resident camp with a subsequent ten month follow-up intervention program. The children participate in a six week day camp where they are engaged in fun-based physical activity and sports, health classes as well as math lessons, Danish language and science classes. All classes are planned and conducted by health professionals and specialist instructors. All physical activity classes are primarily held using outdoor recreational facilities such as soccer fields, basketball courts, and forest areas within bicycling distance to the camp. Three hours of physical activity and sports are scheduled every day, and the classes are designed to reinforce motor skills, fitness, muscle strength, and confidence within the sporting environment. The planned sports activities are both competitive and non-competitive providing the children with both positive experiences in relation to physical activity and tools to cope with competitive situations in their normal environment including commuter bicycling. Bicycles are available for all children. Beside scheduled physical activity the children are encouraged to stay physically active during breaks and leisure time. Six hours a week health classes with the purpose of increasing their knowledge on health issues such as the benefits of a healthy diet and sports participation and increasing body awareness are scheduled. The classes consist of nutritional training, physiology, exercise and goal setting. For this purpose "Appreciative Inquiry" (AI) is used. Briefly, this deals with inquiry into and dialogue about strengths, successes, values, hopes and dreams related to lifestyle behaviors.

The nutritional education consists of theoretical education in the national Danish dietary recommendations in combination with personal guidance at every meal. At the camp food intake is prepared and served according to the national Danish dietary recommendations.(15) The actual eating situation is supervised and guided by specialist instructors, but no calorie restriction is enforced. All camp staff will receive extensive training by specialist instructors with in the field of pedagogic and psychology.

Intervention arm specifications:

Children allocated to this intervention arm will stay at a day camp from 7 a.m. to 8.30 p.m. seven days a week during six weeks including transportation to the day camp. The children will stay at home with their parents outside this time period. The camp is located in the city of Odense, Denmark. The children, together with their family, participate in an initial counseling session. The aim is to support the participants in their efforts to uphold the designed program on diet and food intake. Following this session, the families sign a so-called commitment contract confirming their continuing involvement. During the intervention, text messages will be sent to the children in order to help them comply with the program, and the parents will receive a handbook on dietary recommendations. The children will commute using bicycles to and from the school camp in combination with parent transportation. The children will commute in smaller groups arranged according to the residential area. Active commuting will be supervised and arranged by the camp instructors. Parent transportation will be coordinated by the camp staff.

Early parent involvement - Intervention and Satellite arm:

In the beginning of the intervention a parent council is founded. Experiences from the resident camp project have revealed a positive influence regarding networking and general parent involvement and support due to the foundation of an active parent council (personal communication).

During the day camp the families are offered a dietary course, led by a dietician, consisting of 3x2 hour meetings. Themes at the course are; Healthy cooking, Grocery Shopping, Healthy Eating Patterns in their every day context and parental influence on physical activity behavior.

The subsequent family-based intervention- Intervention and Satellite arm:

After the six week intervention, a family based intervention consisting of four meetings will be planned with the family (the participant and their parents/legal guardian) targeting physical activity and dietary behavior delivered by school health nurses and teachers from the day camp intervention. The following four themes will be attended during the four meetings: "Everyday diet for the family", "Active transport and sports participation", "Weight management in the family" and "Networking and support". Appreciative Inquiry (AI) will be used as a method to equip families with a method to handle challenges related to the targeted behaviors. At all meetings the families will discuss and share experiences related to the central topic of the meeting. The children must be accompanied by at least one parent or legal guardian during the meetings. The investigators have had promising results and feedback from children and families as regards using AI during the family based intervention in the pilot study.

Intervention type 2- control group: Standard intervention:

Children allocated to this intervention will receive a standard intervention, which consist of: 1) one weekly physical activity session (one hour duration) for six weeks arranged by the municipality; 2) two educational sessions, delivered by a dietician and physical activity specialist, for the parents concerning diet and physical activity behavior.

ELIGIBILITY:
Inclusion Criteria:

* Children in the municipality of Odense, Denmark
* Overweight or obese (BMI) according to the International Obesity Task Force

Exclusion Criteria:

* Children who are participating in other research based intervention programmes related to risk factors of heart diseases.
* Children who are following a special school programme.
* Use of weight reducing medicine within 3 months before the baseline measurements
* Children with a motor skill determined handicap of such complexity that it hinders them from participating in the intervention.

Ages: 10 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 115 (Actual)
Dates: Start 2012-04; Primary Completion 2014-07 (Actual); Study Completion 2021-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Lars Bo Andersen, Professor, Principal Investigator — Center of Research in Childhood Health (RICH), University of Southern Denmark
Locations (2):
- Denmark (2):
  - Odense University Hospital, Odense, Funen
  - University of Southern Denmark, Odense, Funen

IPD SHARING:
Plan to Share IPD: Yes
Data is available on request from The Danish National Archives (http://dda.dk/catalogue/30519) after August 2016.
Time Frame: After August 2016
Access Criteria: 1. Data can only be used for scientific and statistical aims and reporting of aggregated information. Not for investigating affairs of private individuals or organisations.
  2. Data can under any circumstances be passed on to a third party, but only be utilized by the user(s) from the project application.
  3. Data can only be used for the purposes stated in the project application for the Danish National Archives.
  4. Considerable changes of the aim will require a new application.
  5. Any publication using the data from the project must bibliographically correct credit the Danish National Archives as well as the principal investigator. Publications must be send to the mailbox og the Danish National Archives attached as a file. The Danish National Archives will forward a copy to the principal investigator.
  6. After utilization of the data it must be deleted or returned to the Danish National Archives.
URL: http://dda.dk/catalogue/30519

REFERENCES:
- [Derived] Thomsen CF, Goharian TS, Larsen KT, Goetze JP, Andersen LB, Jeppesen JL. Intensive Lifestyle Intervention Increases Plasma Midregional Proatrial Natriuretic Peptide Concentrations in Overweight Children. J Am Heart Assoc. 2021 Jul 6;10(13):e020676. doi: 10.1161/JAHA.121.020676. Epub 2021 Jun 28. PMID 34180245
- [Derived] Larsen KT, Huang T, Larsen LR, Olesen LG, Andersen LB, Moller NC. The effect of a multi-component camp-based weight-loss program on children's motor skills and physical fitness: a randomized controlled trial. BMC Pediatr. 2016 Jul 15;16:91. doi: 10.1186/s12887-016-0627-5. PMID 27416906
- [Derived] Larsen KT, Huang T, Moller NC, Andersen LB, Ried-Larsen M. Effectiveness of a one-year multi-component day-camp intervention for overweight children: study protocol of the Odense overweight intervention study (OOIS). BMC Public Health. 2014 Apr 5;14:313. doi: 10.1186/1471-2458-14-313. PMID 24708676
- See also: Institute of Sports Science and Clinical Biomechanics, University of Southern Denmark — http://www.sdu.dk/om_sdu/institutter_centre/iob_idraet_og_biomekanik

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Due to practical circumstances, it was not possible to conduct baseline measurements before randomization. Consequently, 9 participants dropped out before baseline measurements toke place.
Groups:
- Intervention Camp: Children's behavior were controlled each week day for six weeks, and participated in three hours of physical activity every day.
  Intervention camp: The children were participating in a 6 week day camp. The camp contained social activities, physical activity training, usual school classes and health education. All meals (healthy food) were consumed during the camp day.
  A subsequent 46 weeks family based intervention took place after the camp was completed.
- Standard Intervention: Standard intervention: The children were offered a weekly 1 hour training and/or activity session during six weeks. This includes one session where the parents also were invited to get information about diet and exercise.
Period: Overall Study
Arm/Group | Intervention Camp | Standard Intervention
Started | 55 (59 participants where randomized, but 4 dropped out prior to baseline measurements.) | 51 (56 participants where randomized, but 5 dropped out prior to baseline measurements.)
Completed | 48 (Participated in the last follow up measurement.) | 38 (Participated in the last follow up measurement.)
Not Completed | 7 | 13
Not completed — Withdrawal by Subject | 6 | 13
Not completed — Injury in non-camp related sport | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Camp | Standard Intervention | Total
Number analyzed (Participants) | 55 | 51 | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.04 (0.38) | 11.95 (0.46) | 12.00 (0.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 30 | 59
  Male | 26 | 21 | 47
Race/Ethnicity, Customized [Number; unit: participants]
  Danish | 34 | 36 | 70
  Non-Danish | 21 | 15 | 36
Region of Enrollment [Number; unit: participants]
  Denmark | 55 | 51 | 106
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — The BMI is calculated as kg/m^2.
  kg/m^2 | 25.00 (2.80) | 24.52 (3.01) | 24.78 (2.89)
Standardized BMI Z-score [Mean (Standard Deviation); unit: Standardized BMI Z-score] — Based on the International Obesity Task Force (IOTF) 2000 definitions of age and sex adjusted weight status (Cole TJ., 2012).
  According to the IOTF-2000 cut points the body mass index (BMI) of 21.22 kg/m2 at age 12.0 corresponds to a BMI of 25 kg/m2 at age 18.0 for males. The corresponding BMI for females is 21.68 at age 12.0.
  An IOTF Z-score from -1.014 to 1.310 corresponds to normal weight for any given age. Values above are indicative of being overweight. Values below are indicative of being underweight.
  Standardized BMI Z-score | 1.64 (0.37) | 1.54 (0.42) | 1.59 (0.40)
Socio-economic status (SES) [Number; unit: participants] — Based on the mothers highest education level. Data were not available for all participants.
  SES level 1 corresponds to basic school no more than 10 years. SES level 2 corresponds to high school or non-university vocational programs. SES level 3 corresponds to college or university degrees.
  participants
    SES level 1 | 15 | 10 | 25
    SES level 2 | 24 | 15 | 39
    SES level 3 | 13 | 22 | 35
Weight status [Number; unit: participants] — Based on the International Obesity Task Force 2000 definitions of age and sex adjusted weight status. The child was initially invited to participate if he/she was overweight or obese at the screening assessments.
  Some participants had lost weight after the screening and before the baseline measurements, which explains why 9 individuals are normal weight at baseline measurements.
  participants
    Normal weight | 3 | 6 | 9
    Overweight | 36 | 31 | 67
    Obese | 16 | 14 | 30
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] — Measured after 10 minutes in a seated position and calm environment.
  mmHg | 106.64 (7.64) | 103.90 (8.52) | 105.35 (8.14)

OUTCOME MEASURES:

1. Primary Outcome: Change in BMI From Baseline to 12 Months Follow up.
Description: Change in Body Mass Index (BMI) for each intervention arm from baseline (4-6 weeks prior to intervention) to 12 months follow up. BMI is defined as kg/m^2.
  Although three measurements have been conducted, we only report the first and last.
Time Frame: Assessed on 2 occasions: 1) Baseline measurements: 4 - 6 weeks before initiation of interventions. 2) 2nd follow up: 52-53 weeks (12 months) after initiation of interventions.
Population: Only children that participated in both the baseline and the follow up measurements were included in the results.
Measure: Mean (95% Confidence Interval); unit: BMI (kg/m^2)
Arm/Group | Intervention Camp | Standard Intervention
Number analyzed (Participants) | 48 | 38
BMI (kg/m^2) | -1.1 [-1.7 to -0.6] | 0.1 [-0.4 to 0.6]

2. Secondary Outcome: Change in Cognitive Function From Baseline to 12 Months Follow up.
Description: To assess cognitive function the following test are used: The Stroop Color and word test; Trail making test (part A and B); Rey complex figure test and recognition trial; Symbol digit modalities Test; Behavior rating inventory of executive function.
Time Frame: as for outcome 1
Reporting Status: Not Posted, anticipated posting 2021-07

3. Secondary Outcome: Change in Motor Skills From Baseline to 12 Months Follow up.
Description: To assess motor skills, the Movement Assesment Battery for Children 2 (Movement ABC-2) test for 11-16 year olds was applied. The battery allows for recording a number of different aspects of a child's movement skills in a systematic way. In this study we only used the quantitative part of the test (it also includes a qualitative part). This includes 3 tests for hand skills (fine motor skills), 2 tests for throwing and catching balls, and 3 tests for balance skills. Each subtest returns a score, which is summarized and then equivalent to a percentile score (based on norm data from a standard population in a table from the Movement ABC-2 compendium). The percentile score is reported as the overall motor skills. The scale is from 0.1 to 99.9 (normal distributed with an average of 50) and higher scores mean better motor skills.
Time Frame: as for outcome 1
Population: Only children that participated in both the baseline and the follow up measurements were included in the results.
Measure: Mean (95% Confidence Interval); unit: Percentile score on a scale
Arm/Group | Intervention Camp | Standard Intervention
Number analyzed (Participants) | 46 | 36
Percentile score on a scale | 6.4 [-0.5 to 13.3] | 22.6 [13.2 to 32.0]

4. Secondary Outcome: Change in Body Composition From Baseline to 12 Months Follow up.
Description: Measurements of fat mass and lean tissue mass using dual-energy X-ray absorptiometry.
Time Frame: as for outcome 1
Population: Only children that participated in both the baseline and the follow up measurements were included in the results. As this test took place on a different time and location than most other tests, the number of participants differs from many other tests.
Measure: Mean (95% Confidence Interval); unit: Change in percent body fat
Arm/Group | Intervention Camp | Standard Intervention
Number analyzed (Participants) | 47 | 39
Change in percent body fat | -3.8 [-5.1 to -2.6] | -2.0 [-3.4 to -0.7]

5. Secondary Outcome: Change From Baseline in Brain-derived Neurotrophic Factor (BDNF) at 12 Months.
Description: The chronic level of serum brain-derived neurotrophic factor (BDNF) is assessed in fasting blood samples.
Time Frame: as for outcome 1
Reporting Status: Not Posted, anticipated posting 2021-07

6. Secondary Outcome: Change From Baseline in Blood Pressure at 12 Months.
Description: Blood pressure will be measured in up-right sitting position after resting supine for ten minutes. A minimum of five measurements will be conducted with one minute intervals.
Time Frame: as for outcome 1
Reporting Status: Not Posted, anticipated posting 2021-07

7. Secondary Outcome: Change From Baseline in Subclinical Atherosclerosis Using B-mode Ultrasound: Carotid Intima Media Thickness and Carotid Elasticity at 12 Months.
Description: The Carotid Intima Media and Carotid Elasticity are measured on 2 sites (posterior and lateral) of the far wall 1 cm proximal to the bifurcation on both sides of the common carotid artery.
Time Frame: as for outcome 1
Reporting Status: Not Posted, anticipated posting 2021-08

8. Secondary Outcome: Change From Baseline in Cardio-respiratory Fitness at 12 Months.
Description: Cardio-respiratory fitness will be assessed using a progressive bicycle ergometer protocol after a 5 minutes warm-up by means of indirect calorimetry (Innovision, Odense, Denmark).
Time Frame: as for outcome 1
Reporting Status: Not Posted, anticipated posting 2021-07

9. Secondary Outcome: Change From Baseline in Insulin Level at 12 Months.
Description: The level of insulin is assessed in fasting blood samples.
Time Frame: as for outcome 1
Reporting Status: Not Posted, anticipated posting 2021-07

10. Secondary Outcome: Change From Baseline in Glucose Level at 12 Months.
Description: The level of glucose is assessed in fasting blood samples.
Time Frame: as for outcome 1
Reporting Status: Not Posted, anticipated posting 2021-07

11. Secondary Outcome: Change From Baseline in Blood Lipids at 12 Months.
Description: The levels of lipids are assessed in fasting blood samples.
Time Frame: as for outcome 1
Reporting Status: Not Posted, anticipated posting 2021-07

12. Secondary Outcome: Change From Baseline in C-Reactive Protein at 12 Months.
Description: The level of c-reactive-protein is assessed in fasting blood samples.
Time Frame: as for outcome 1
Reporting Status: Not Posted, anticipated posting 2021-07

13. Secondary Outcome: Change From Baseline in Waist/Hip Circumference at 12 Months.
Description: Hip circumference will be measured at the level of the great trochanter. Waist circumference will be measured between the lower costal margin and the iliac crest.
Time Frame: as for outcome 1
Reporting Status: Not Posted, anticipated posting 2021-07

14. Secondary Outcome: Change in Clustered Cardiovascular Disease (CVD) Risk Factor
Description: The CVD risk factor is the mutual presence of five different health outcomes based on the Metabolic Syndrome. It is calculated by creating a composite risk score (mean of z-scores) of: 1) Insulin resistance (Homeostatic Model Assessment for Insulin Resistance (HOMA-IR)), 2) Systolic blood pressure, 3) triglyceride, 4) total cholesterol/HDL ratio, 5) Abdominal fatness (by Dual-energy X-ray absorptiometry (DXA)), and 6) aerobic fitness.
Time Frame: as for outcome 1
Reporting Status: Not Posted, anticipated posting 2021-07

15. Secondary Outcome: Change From Baseline in Physical Strength at 12 Months.
Description: Will be measured by hand grip and Sargent vertical jump.
Time Frame: as for outcome 1
Reporting Status: Not Posted, anticipated posting 2021-07

ADVERSE EVENTS:
Time Frame: During the 48 weeks following the intervention. Monitoring were non-systematic.
Description: Health professionals (school nurses) met families that choose to participate in the following meetings throughout the 48 weeks following the intervention. If any of the children showed signs of eating disorders or self harm, they would react appropriately. The screening were non-systematic.
Groups:
- Camp Intervention: The intervention camp consisted of a six-week multi-component day camp including increased physical activity, healthy diet and health education followed by 46 weeks of family-based habitual intervention.
  The standard care arm was offered two weekly hours of physical activity training for six weeks.
- Standard Internvention: In the Standard intervention children were offered a weekly 1-hour training and/or activity session during six weeks. This includes one session where the parents also were invited to get information about diet and exercise.
Arm/Group | Camp Intervention | Standard Internvention
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/51
Other Adverse Events (participants affected / at risk) | 0/55 | 0/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Camp Intervention (N=55) | Standard Internvention (N=51)
Eating disorder (Psychiatric disorders) | 0 (0) | 0 (0) — School nurses were observant, although in a non-systematic manner, whether any of the children showed signs of eating disorder during the 48 week family-based intervention period.
Self harm (Psychiatric disorders) | 0 (0) | 0 (0) — School nurses were observant, although in a non-systematic manner, whether any of the children showed signs of self harm during the 48 week family-based intervention period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No